CLINICAL TRIAL: NCT05102695
Title: Study of CRP, Ferritine and D-Dimer in Covid-19 Patients Admitted To Respiratory ICU in Assuit University Hospitals
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mina Ibraheem Anis, Resident Doctor at chest department assuit university, Assiut University
Other Study IDs: CRP, Ferritine,d-dimer
Record Dates: First submitted 2021-10-28; First posted 2021-11-01 (Actual); Last update posted 2021-11-05 (Actual); Status verified 2021-10

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Serum CRP , ferritine and d-dimer — Correlation between the results of the tests with outcome of the patient

SUMMARY:
To Study serum CRP, D-dimer and serum ferritin in adult patients with COVID-19 for the presence or absence of clinically validated definitions of mortality, severe COVID-19, ARDS, and intensive care unit (ICU) care.

DETAILED DESCRIPTION:
Inflammatory markers are often elevated in patients with COVID-19, notably C-reactive protein (CRP), D-dimer, lactate dehydrogenase (LDH), IL-6and ferritin. Multiple prior studies have found correlations between various biomarkers and clinical outcomes in patients with COVID-19 However, the clinical utility of these various biomarkers for risk-stratification and determining prognosis among patients with COVID-19 is evolving and still ill-defined [4] C-reactive protein (CRP) is an acute inflammatory protein that increases up to 1,000-fold at sites of infection or inflammation. CRP is produced as a homopentameric protein, termed native CRP (nCRP), which can irreversibly dissociate at sites of inflammation and infection into five separate monomers, termed monomeric CRP (mCRP). CRP is synthesized primarily in liver hepatocytes but also by smooth muscle cells, macrophages, endothelial cells, lymphocyte. CRP showed different distribution feature and existed differences in various ages, clinical types and outcomes of COVID-19 patients. The features corresponded with disease progression [5] There is an over-exuberant cytokine release with hyperferritinemia leading to the idea that COVID-19 is part of the hyperferritinemic syndrome spectrum. Indeed, very high levels of ferritin can occur in other diseases including hemophagocytic lymphohistiocytosis, macrophage activation syndrome, adult-onset Still's disease, catastrophic antiphospholipid syndrome and septic shock. Numerous studies have demonstrated the immunomodulatory effects of ferritin and its association with mortality and sustained inflammatory process. High levels of free iron are harmful in tissues, especially through the redox damage that can lead to fibrosis. Iron chelation represents a pillar in the treatment of iron overload. In addition, it was proven to have an anti-viral and anti-fibrotic activity. Through analysis of the pathogenic role of iron during SARS-CoV-2 infection so, iron depletion therapy may be a novel therapeutic approach in the COVID-19 pandemic.[6] Cytokine storm is an interesting point in COVID-19 patients. High levels of inflammatory cytokines were observed in COVID-19 patients with more severe disease and were associated with pulmonary inflammation, lung damage and multiple organ failure. IL-6 is an important cytokine whose production is related with various inflammatory diseases. Subjects with SARS-CoV-2 had high levels of IL-6 that were correlated with patient symptomatology including pulmonary inflammation and extensive lung damage. Additionally, patients with SARS-CoV-2 infection had low levels of suppressor of cytokine signaling-3, which regulates and stimulates the negative feedback mechanism of IL-6. On the same line, another study reported that IL-6 levels were higher in severe COVID-19 patients and this may be used as one of the bases for predicting the transition from mild to severe infection. Some studies showed that COVID-19 patients in intensive care had lower CD8+ T cell counts and their total CD4+ and CD8+ T cell counts were also negatively correlated with TNF-α and IL-6 concentrations. In addition, recent studies showed that higher level of IL-6, CRP and also IL-10 were more significant rather than other cytokines in critical group of COVID-19 patients. It can be suggested that immune dysregulation is a highly important point and therapeutic target for COVID-19 patients. The reasons for the large scale of the inflammatory cytokines are not clear, but it could play a crucial role in cell apoptosis associated with organ damage.[7] Some studies have reported that the humanized monoclonal antibody against IL-6 receptors, tocilizumab, can be used in COVID-19 treatment based on its cytokine storm blocking property. A recent Chinese retrospective study showed that tocilizumab improved fever, CRP levels and hypoxemia without leading to any significant adverse reactions in 21 severe COVID-19 patients. According to the Italian guidelines, tocilizumab can only be used for COVID-19 patients who are at the end of the high viral load phase, with interstitial pneumonia, heavy respiratory insufficiency and high lL-6 and/or D-dimer/CRP/ferritin/fibrinogen levels [8] D-dimer is a degradation product of crosslinked fibrin resulting from plasmin cleavage. During fibrinolysis plasmin may degrade fibrin monomers, crosslinked fibrin polymers and possibly fibrinogen during systemic fibrinolysis following alpha2 depletion. All these fragments are collectively called fibrin degradation products (FDPs). D-dimer constitutes two adjacent fibrin 'D' domains (ends) that are cross-linked and released as an intact fragment, hence the name D-dimer. Several studies from Wuhan have shown elevated D-dimer in COVID-19 patients is associated with higher mortality, Although it is not clear what effect anticoagulation has on D-dimer levels in the setting of COVID-19, very low D-dimer levels are usually observed in patients receiving anticoagulation.Because D-dimer is a product of cross-linked fibrin, it is considered a sensitive biomarker to rule out venous thromboembolism. However, D-dimer has low specificity as there are many other conditions with ongoing activation of the hemostatic system in which D-dimer can be elevated such pregnancy, inflammation, malignancy, trauma, liver disease (decreased clearance), heart disease, sepsis or as a result of hemodialysis, CPR or recent surgery.[9] Although several studies have suggested that severe disease may be associated with elevated CRP, Ferritine and D-Dimer, the results across these studies are not entirely consistent. So far, it is unclear whether inflammatory markers are significantly higher in patients with severe COVID-19 than in those with mild disease.[10] So the investigators will try to assess CRP, Ferritine and D-Dimer and their association with the severity of the COVID-19 disease.

ELIGIBILITY:
Inclusion Criteria:

* -Cases aged 18 years and over. -Cases diagnosed as COVID-19 by radiology or with positive PCR. -Cases admitted to Assuit University Hospitals.

Exclusion Criteria:

* -Cases less than 18 Years old. -Cases Diagnosed as COVID-19 and Discharged from emergency department for home isolation. -Cases who refused the use of their data.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Covid-19 poaitive patients admitted to assuit unirversity hospitals
Sampling Method: Non-Probability Sample
Enrollment: 160 (Estimated)
Dates: Start 2022-01-01 (Estimated); Primary Completion 2023-03-01 (Estimated); Study Completion 2023-04-01 (Estimated)

PRIMARY OUTCOMES:
Correlation between results and outcome of the patients | Baseline
  Either severe infection , ICU admission or death with CRP > 23 mg\L or < 10 mg\ L , Ferritine > 440 ng\ml or < 300 ng\ml or D-dimer. > or < .9 mg\L